CLINICAL TRIAL: NCT05671705
Title: Effect of Sarcopenia in Stroke Patients
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Collaborators: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Sun Im, MD., PhD., The Catholic University of Korea
Other Study IDs: VC22ONDI0185
Record Dates: First submitted 2022-11-24; First posted 2023-01-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Sarcopenia
MeSH Terms: conditions — Stroke; Sarcopenia | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stroke patients with sarcopenia: Group will be stratified according to gender
  Interventions: Diagnostic Test: DEXA Scan
- Stroke patients without sarcopenia: Group will be stratified according to gender
  Interventions: Diagnostic Test: DEXA Scan

INTERVENTIONS:
Diagnostic Test: DEXA Scan — Fu of diagnostic tests
  Other Names: Serum biomarkers, SEMG signals and MRI changes

SUMMARY:
Primary research purpose:

-Prospective study to screen post stroke patients with sarcopenia and evaluate its effect on recovery

Secondary research purpose:

* To determine the degree of sarcopenia and correlation with poor functional prognosis of stroke in the stroke patient group.
* To determine the degree of sarcopenia and correlation with dixon MRI of thigh muscle
* To evaluate surface EMG (SEMG)-based signals and correlation with sarcopenia
* To determine the degree of sarcopenia and correlation with brain morphometric changes

DETAILED DESCRIPTION:
Patients with first-ever stroke will be enrolled and assessed for sarcopenia. The evaluation parameters will include standard sarcopenia parameters and also SEMG-based signals and imaging studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years of age or older, stroke patients with first onset within 4 weeks

Exclusion Criteria:

* Patients who have not been evaluated for sarcopenia
* Patients with neuromuscular diseases other than stroke that may affect gait function
* Patients unable to conduct clinical trials according to instructions
* Patients with uncontrolled medical/surgical disease
* Patients with metal substances in the body such as cardiac pacemakers, cochlear implants, etc.
* Patients who have difficulty collecting blood
* Patients who are difficult to follow up after 6 months of onset due to moving to another area
* Patients who have Parkinson's disease, dementia, or have a history of neuromuscular diseases such as Guillain-Barré syndrome or myasthenia gravis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Recruited subjects will be allocated into 4 different groups according to presence of sarcopenia according to the Asian Working Group for Sarcopenia (2019) criteria.
  * Post stroke male patients with sarcopenia
  * Post stroke female patients with sarcopenia
  * Post stroke male patients without sarcopenia
  * Post stroke female patients without sarcopenia
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Change of Modified Rankin Scale | 6 months from the first onset of the stroke
  Functional Disability -> The scale runs from 0-6, running from perfect health without symptoms(0) to death(6).

SECONDARY OUTCOMES:
Hand grip strength | within 4 weeks, 4 weeks, 8 weeks, 6 months from the first onset of the stroke
  Grip strength: Grip strength will be measured using a dynamometer
quadriceps muscle strength | within 4 weeks, 4 weeks, 8 weeks, 6 months from the first onset of the stroke
  Lower extremity strength assessment:change in isometric quadriceps muscle strength (kg) from initial evaluation to the final evaluation
Fugl-Meyer motor scale | within 4 weeks, 4 weeks, 8 weeks, 6 months from the first onset of the stroke
  Motor function assessment : Fugl-Meyer motor scale from initial evaluation to the final evaluation (Upper Extremity maximum score = 66; Lower Extremity maximum score = 34, Higher score means better outcome)
Functional Ambulation Category | within 4 weeks, 4 weeks, 8 weeks, 6 months from the first onset of the stroke
  Gait function assessment : Functional Ambulation Category from initial evaluation to the final evaluation (Minimum 0, Maximum 5; Higher score means better outcome)
Berg balance scale | within 4 weeks, 4 weeks, 8 weeks, 6 months from the first onset of the stroke
  Balance function: change in Berg balance scale from initial evaluation to the final evaluation (Minimum score 0, Maximum score 56, Higher score means better outcome)
Brain MRI | within 4 weeks and 6 months from the first onset of the stroke
  Brain atrophy : change in the Global cortical atrophy scale(0-3) of the cerebral cortex from initial evaluation to the final evaluation
Thigh Dixon MRI | within 4 weeks and 6 months from the first onset of the stroke
  Muscle quality : muscle circumference measured by the thigh MRI from initial evaluation to the final evaluation
Muscle ultrasonography | within 4 weeks and 6 months from the first onset of the stroke
  muscle thickness(cm) measured by the ultrasound of the quadriceps muscle from initial evaluation to the final evaluation
serum biomarkers for sarcopenia | within 4 weeks from the first onset of the stroke
  BNDF, IL-6
Digitalized SEMG signals | within 4 weeks, 4 weeks, 8 weeks, 6 months from the first onset of the stroke
  state of the art EMG signals will be collected to assess muscle quality changes after stroke

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - The Catholic University of Korea, Bucheon-si, Gyeonggi-do
  - St. Vincent's Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Undecided